CLINICAL TRIAL: NCT01171833
Title: Effect of Ventilation on Speed of Induction of Anesthesia in Desflurane, Sevoflurane, and Isoflurane
Brief Title: Ventilatory Effect on Speed of Anesthesia Under Various Inhaled Anesthetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Junyong In, Assistant professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: J In 2010-1
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Pharmacokinetics of Inhaled Anesthetics
Keywords: Anesthetic induction; Desflurane; Isoflurane; Sevoflurane; Ventilation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Sevoflurane; Desflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A(Sevoflurane) (Experimental): Twelve patients will be enrolled in this group. They will be divided into subgroups with ventilatory settings.
  Each subgroup has 4 patients.
  A8: tidal volume(8 ml/kg) and respiratory rate(10 /min) A10: tidal volume(10 ml/kg) and respiratory rate(10 /min) A12: tidal volume(12 ml/kg) and respiratory rate(10 /min)
  Interventions: Drug: Sevoflurane
- Group B(Desflurane) (Experimental): Twelve patients will be enrolled in this group. They will be divided into subgroups with ventilatory settings.
  Each subgroup has 4 patients.
  A8: tidal volume(8 ml/kg) and respiratory rate(10 /min) A10: tidal volume(10 ml/kg) and respiratory rate(10 /min) A12: tidal volume(12 ml/kg) and respiratory rate(10 /min)
  Interventions: Drug: Desflurane
- Group C(Isoflurane) (Experimental): Twelve patients will be enrolled in this group. They will be divided into subgroups with ventilatory settings.
  Each subgroup has 4 patients.
  A8: tidal volume(8 ml/kg) and respiratory rate(10 /min) A10: tidal volume(10 ml/kg) and respiratory rate(10 /min) A12: tidal volume(12 ml/kg) and respiratory rate(10 /min)
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Sevoflurane — 2.0 vol% prefilled in a corrugated circuit.
  Other Names: Sevorane
  Arms: Group A(Sevoflurane)
Drug: Desflurane — 6.0 vol% prefilled in a corrugated circuit.
  Other Names: Suprane
  Arms: Group B(Desflurane)
Drug: Isoflurane — 1.2 vol% prefilled in a corrugated circuit.
  Other Names: Aerane
  Arms: Group C(Isoflurane)

SUMMARY:
Three groups of patients are going to have minor surgery under general anesthesia with inhaled anesthetics and different ventilatory setting (Tidal volume: 8, 10, 12 ml/kg, respiratory rate: 10/min each). Group A (Sevoflurane) will use sevoflurane, group B (Desflurane) will use desflurane, and group C (Isoflurane) will use isoflurane. It will be observed differences among the groups for ventilatory effects on speed of induction.

Duration of this randomised controlled trial will be about 3 months. Estimated sample size will be 36 patients(12 in each group).

DETAILED DESCRIPTION:
No premedicant will be given. The anesthetic workstation and a circulatory circuit will be prefilled with 1.0 MAC of inhaled anesthetic that will be selected randomly.

* Group A (n=12): Sevoflurane 2.0 vol%
* Group B (n=12): Desflurane 6.0 vol%
* Group C (n=12): Isoflurane 1.2 vol%

Each group has 3 subgroups according to the ventilatory setting that will also be randomly determined.

* Hypoventilation: tidal volume 8 ml/kg, respiratory rate 10 /min
* Normoventilation: tidal volume 10 ml/kg, respiratory rate 10 /min
* Hyperventilation: tidal volume 12 ml/kg, respiratory rate 10 /min

Patients will be preoxygenated with 100% oxygen (5 L/min) for 5 minutes under pulse oximeter, EKG, and noninvasive blood pressure monitoring. Bispectral index (BIS) monitor will be applied.

The induction of general anesthesia will start with propofol (2 mg/kg), rocuronium (0.8 mg/kg) and remifentanil infusion (0.1 mcg/kg/min). The size of a tracheal tube will be 7.5 mm (ID) for male, 7.0 mm (ID) for female. After intubation, anesthesia workstation will be connected to the tracheal tube. Ventilation will start, and that point will be time 0. During 720 seconds, inspiratory (PIgas) and end-tidal concentration of inhaled anesthetics (ETgas), end-tidal partial pressure of carbon dioxide, and BIS will be measured at time 0, 30, 60, 90, 120 ,150, 180, 240, 300, 360, 480, 600, and 720 seconds. Mean blood pressure and heart rate will also be recorded every 2 minutes. Fresh gas flow will be kept at 6 L/min with 100% oxygen.

The fraction of ETgas/PIgas will be analyzed with nonlinear mixed effects modeling.

Estimated sample size will be 36 patients (12 in each group, 4 in each ventilatory settings).

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I, II
* Age: 20-60 years male and female
* Elective schedule with minor surgery
* BMI < 30

Exclusion Criteria:

* Patients with pulmonary, cardiac, endocrinal, neuromuscular and neurological diseases or past history
* Upper airway anomaly or deformity
* ASA PS III or higher
* Pregnant women
* BMI >= 30

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
End-tidal concentrations of isoflurane, sevoflurane and desflurane, and BIS values with hypo-, normo-, hyperventilation | at 0, 30, 60, 90, 120, 180, 240, 300, 360, 480, 600, 720 sec after volatile gas starts
  The inspiratory, and end-tidal concentrations of volatile anesthetics, partial pressure of end-tidal carbon dioxide will be recorded from an S/5 Avance anesthetic workstation (Datex-Ohmeda) and an embedded monitor. BIS values are measured with a BIS monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Junyong In, MD, Principal Investigator — Dept. of anesthesiology and pain medicine, Dongguk University Ilsan Hospital